CLINICAL TRIAL: NCT04169009
Title: Persistence of Protection Conferred by Shingrix Against Herpes Zoster
Brief Title: Persistence of Protection by Shingrix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-0580; 1U01AI141919-01 (NIH)
Record Dates: First submitted 2019-09-25; First posted 2019-11-19 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Herpes Zoster
Keywords: immunology
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ZVL >5 years previously (Active Comparator): Participants have received Zostavax (ZVL) at least 5 years previously. Will be administered intradermal vOka varicella zoster virus (ZVL) in non-dominant deltoid. A skin biopsy will be performed at the injection site on 20 subjects.
  Interventions: Biological: Zostavax
- ZVL 6-12 months previously (Active Comparator): Participants who received ZVL 6-12 months previously will be administered an intradermal dose of vOka varicella zoster virus (ZVL) in non-dominant deltoid.
  Interventions: Biological: Zostavax
- No previous ZVL (Active Comparator): Participants who've never received a shingles vaccine will be given the 2 standard doses of RZV. Six months later they will be given the intradermal dose of vOka varicella zoster virus (ZVL) in the non-dominant deltoid.
  Interventions: Biological: Zostavax; Biological: Shingrix
- SRX >5 years previously (Active Comparator): Participants have received Shingrix at least 5 years previously. Will be administered intradermal vOka varicella zoster virus (ZVL) in non-dominant deltoid. A skin biopsy will be performed at the injection site on 20 subjects.
  Interventions: Biological: Zostavax

INTERVENTIONS:
Biological: Zostavax — Intradermal injection of Zostavax
Biological: Shingrix — Given to subjects in Arm 4 who've never had a herpes zoster vaccine
  Arms: No previous ZVL

SUMMARY:
The study plans to learn more about how the shingles vaccine, Shingrix (SRX), successfully prevents shingles in older people. Two vaccines are currently approved by the Food and Drug Administration (FDA) to prevent shingles. Zostavax is a live virus vaccine which has been available since 2006 and prevents shingles about 50% of the time, though it is less effective the older a person is when they receive it. Shingrix, which was approved by the FDA in 2017, is not a live virus, but has an additive in the vaccine to boost immune response. It is about 97% effective at preventing shingles regardless of a person's age and so far has been effective for at least 4 years after vaccination. Because Zostavax has live virus in it, giving a "challenge" dose of Zostavax - vOka varicella zoster virus - to people who have received both vaccines (Zostavax or Shingrix) in the past, will allow researchers to learn more about how the body works to prevent shingles and how any shingles vaccination helps protect against shingles.

DETAILED DESCRIPTION:
The primary endpoint of this study was the area under the concentration/time curve of quantitative VZV DNA in plasma. However, all the VZV DNA measurements were below the lower limit of quantitation of the assay. Due to this unexpected outcome, we performed a qualitative analysis of presence or absence of VZV DNA in plasma at Day ≥3 after the vOka challenge.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-85
* General good health
* Women of non-childbearing potential must be postmenopausal or have undergone hysterectomy or bilateral oophorectomy
* ARM 1 ONLY: Documented evidence of immunization with ZVL or SRX at least 5 years previously
* ARM 2 ONLY; Documented evidence of immunization with ZVL 6-12 months prior to enrollment
* ARM 3 ONLY: Have never received any shingles vaccination

Exclusion Criteria:

* Prior history of herpes zoster (HZ)
* Blood products received in the 3 months prior to study enrollment or planned for the subsequent week for Arm 1; Arm 2 requires same exclusion; Arm 3 extends the exclusion to the week after the vOka challenge, which is 6 months after completing SRX administration.
* Significant immune suppressive illness or therapy
* Concomitant vaccine received within 2 (inactive) or 4 (live) weeks prior to the study or during the first week of the study.
* Women of childbearing potential.
* Pregnancy or breastfeeding.
* Participation in a concurrent clinical study in which the subject will be exposed to and investigational product during the period starting 7 days before the first dose of study vaccine through the completion of the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Weinberg, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Clinical Trials Center at University of Colorado Anschutz Medical Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ZVL >5 Years Previously (Cohort 1): Participants have received Zostavax (ZVL) at least 5 years previously. Will be administered intradermal vOka varicella zoster virus (ZVL) in non-dominant deltoid. A skin biopsy will be performed at the injection site on 20 subjects.
  Zostavax: Intradermal injection of Zostavax
- ZVL 6-12 Months Previously (Cohort 3): Participants who received ZVL 6-12 months previously will be administered an intradermal dose of vOka varicella zoster virus (ZVL) in non-dominant deltoid.
  Zostavax: Intradermal injection of Zostavax
- No Previous ZVL (Cohort 4: Participants who've never received a shingles vaccine will be given the 2 standard doses of RZV. Six months later they will be given the intradermal dose of vOka varicella zoster virus (ZVL) in the non-dominant deltoid.
  Zostavax: Intradermal injection of Zostavax
  Shingrix: Given to subjects in Arm 4 who've never had a herpes zoster vaccine
- SRX >5 Years Previously (Cohort 2): Participants have received Shingrix at least 5 years previously. Will be administered intradermal vOka varicella zoster virus (ZVL) in non-dominant deltoid. A skin biopsy will be performed at the injection site on 20 subjects.
  Zostavax: Intradermal injection of Zostavax
Period: Overall Study
Arm/Group | ZVL >5 Years Previously (Cohort 1) | ZVL 6-12 Months Previously (Cohort 3) | No Previous ZVL (Cohort 4 | SRX >5 Years Previously (Cohort 2)
Started | 18 | 32 | 35 | 20
Completed | 18 | 31 | 35 | 19
Not Completed | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZVL >5 Years Previously (Cohort 1) | ZVL 6-12 Months Previously (Cohort 3) | No Previous ZVL (Cohort 4 | SRX >5 Years Previously (Cohort 2) | Total
Number analyzed (Participants) | 18 | 32 | 35 | 20 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 30 | 28 | 9 | 78
  >=65 years | 7 | 2 | 7 | 11 | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.14 [59.44 to 75.56] | 56.37 [54.31 to 60.48] | 61.15 [57.82 to 63.44] | 67.79 [61.09 to 78.35] | 60.74 [57.43 to 65.16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 25 | 12 | 66
  Male | 4 | 17 | 10 | 8 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 16 | 25 | 33 | 18 | 92
  Non-Hispanic Black | 1 | 5 | 1 | 1 | 8
  Hispanic | 0 | 1 | 0 | 0 | 1
  Other | 1 | 1 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 18 | 32 | 35 | 20 | 104

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Varicella-Zoster Virus (VZV) DNAemia
Description: Varicella-Zoster Virus (VZV) DNAemia will be measured by polymerase chain reaction (PCR) as a surrogate for viremia over the first 7 days after vOka intradermal (ID) challenge. The outcome measure will be the area under the concentration time curve of the VZV DNAemia expressed in DNA copies/ml of blood.
Time Frame: Until VZV DNA is undetectable in the blood, measured up to Day 7
Measure: Geometric Mean (Standard Deviation); unit: DNA copies per/mL
Arm/Group | ZVL >5 Years Previously (Cohort 1) | ZVL 6-12 Months Previously (Cohort 3) | No Previous ZVL (Cohort 4 | SRX >5 Years Previously (Cohort 2)
Number analyzed (Participants) | 18 | 32 | 35 | 20
DNA copies per/mL | NA (NA) — Viral load below lloq (lower limit of quantification) | NA (NA) — Viral load below lloq (lower limit of quantification) | NA (NA) — Viral load below lloq (lower limit of quantification) | NA (NA) — Viral load below lloq (lower limit of quantification)

ADVERSE EVENTS:
Time Frame: AEs starting within 7 days after injection and Grade ≥ 3 will be recorded and followed until resolution. ZVL - Subjects in Cohort 3 receiving ZVL on Day 0 will be followed for AEs for 7 days. RZV - Subjects in Cohort 4 receiving RZV on Day 0 and Day 60 will also be followed for AEs for 7 days after each injection. Any Grade ≥ 3 will be recorded and followed until resolution. All study procedure AEs will be followed until resolution.
Groups:
- No Previous ZVL (Cohort 4): Participants who've never received a shingles vaccine will be given the 2 standard doses of RZV. Six months later they will be given the intradermal dose of vOka varicella zoster virus (ZVL) in the non-dominant deltoid.
  Zostavax: Intradermal injection of Zostavax
  Shingrix: Given to subjects in Arm 4 who've never had a herpes zoster vaccine
Arm/Group | ZVL >5 Years Previously (Cohort 1) | ZVL 6-12 Months Previously (Cohort 3) | No Previous ZVL (Cohort 4) | SRX >5 Years Previously (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/32 | 0/35 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/32 | 0/35 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/32 | 16/35 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZVL >5 Years Previously (Cohort 1) (N=18) | ZVL 6-12 Months Previously (Cohort 3) (N=32) | No Previous ZVL (Cohort 4) (N=35) | SRX >5 Years Previously (Cohort 2) (N=20)
Body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) — Generalized body aches
shaking chills (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
decreased range of motion LUE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dizziness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — 103.5 F
Worsening back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
felt feverish (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT04169009/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT04169009/ICF_001.pdf